CLINICAL TRIAL: NCT03058172
Title: Study of Olfaction / Vision Interactions in Expert and Novice Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0685
Record Dates: First submitted 2017-02-08; First posted 2017-02-20 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Odors (food and non-food) (Other): Odorants diluted in mineral oil.
  Interventions: Other: Odor presentation (for participants' perception)
- Pictures (food and non-food) (Other): Pictures of objects or scenes.
  Interventions: Other: Image presentation (for participants' perception)

INTERVENTIONS:
Other: Odor presentation (for participants' perception) — Several different odors will be diffused by an olfactometer under the participants' nostrils, though a controlled airflow, and synchronously with the participants' respiration. fMRI designs require repeated stimulus presentation. Odors will also be presented (in flasks or in odor pens) outside the scanner.
  Arms: Odors (food and non-food)
Other: Image presentation (for participants' perception) — Several different pictures will be displayed in front of the participants' face, though a through a mirror system in the scanner, or on a computer screen outside the scanner.
  Arms: Pictures (food and non-food)

SUMMARY:
The aim of this research project is to better understand the reciprocal influence of visual and olfactory systems on cerebral activity evoked by odors and visual stimuli. Given the importance of olfacto-visual learning in expert situations, the degree of expertise in olfaction will also be considered. In addition, the investigators will try to better understand the differences between expert and non-expert populations in olfaction through different levels of approach: sensory, genetic and cerebral. To achieve this, the investigators will use psychophysical tests, genetic analyzes and a non-invasive technique, functional magnetic resonance imaging (fMRI) to measure the brain activity of human subjects - novices or experts in olfaction - in response to different visual and olfactory stimuli.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* men and women, aged 18-85 years old
* subjects with social security cover
* expertise in olfaction for half of the subjects (60)

Exclusion Criteria:

* subjects younger than 18 and older than 85
* subjects with contraindications to fMRI, i.e. with pacemaker / insulin pump / metal prosthesis / intracerebral clip / neurosensory stimulator / implantable defibrillator / cochlear implants / ferromagnetic ocular or cerebral foreign body close to the nerve structures / ventriculoperitoneal neurosurgical bypass valves / braces and other non-removable metallic dental device / claustrophobic, non-cooperating or agitated subjects.
* pregnant or breastfeeding women
* subjects with known olfactory disorder
* subjects with known neurological disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04-15 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Brain activity | During the 2-hour testing session (one session per participant)
  fMRI 3T scanner in CERMEP imaging center (Bron - see web link at the end of the document), allowing anatomical measures, connectivity between olfactory and other regions (DTI), activation pattern in olfactory and visual areas.

SECONDARY OUTCOMES:
Genotyping | Sampling during the 2-hour testing session (one session per participant), analyses within 6 years after sampling
  Genotyping from saliva samples by AMIS laboratory or a genotyping platform in Toulouse or Evry (see web links at the end of the document)
Olfactory abilities | During the 2-hour testing session (one session per participant)
  Threshold detection, discrimination between odorants and odor identification, measured with standardized olfactory tests
Perception | During the 2-hour testing session (one session per participant)
  Assesment of the perceptual profile of the stimulus on visual analogue scale (verbal report of how the olfactory/visual stimulus is perceived).
Response times | During the 2-hour testing session (one session per participant)
  Response time to the olfactory/visual stimulus in millisecond

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric FAURE, MD, Principal Investigator — Infirmerie Protestante
Locations (1):
- Infirmerie Protestante, Caluire-et-Cuire, France